CLINICAL TRIAL: NCT03150537
Title: Comparison of Routine IM Influenza Immunization and Administration by Jet-injector (Med-Jet MIT H4™ & Disposable Cartridge) in Healthy Young Adults
Brief Title: Comparison of Routine IM Influenza Immunization and Administration by Jet-injector (Med-Jet H4™) in Healthy Young Adults
Acronym: Med-Jet H4™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: brian.ward (Other)
Collaborators: MEDICAL INTERNATIONAL TECHNOLOGIES (MIT CANADA) INC. (Unknown); MedTeq (Industry)
Responsible Party: Sponsor-Investigator, brian.ward, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: RI-MUHC: 2017-3307
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Needle Phobia
Keywords: jet injector; influenza vaccine; immune response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Eighty healthy adults (18-49 years of age) will be randomized 1:1 to receive:
  * A single dose of trivalent inactivated influenza vaccine (TIV: Fluviral™: 0.5mL IM)
    * Half will receive the vaccine using a pre-filled syringe
    * Half will receive the vaccine using a multi-dose vial
  * Or,the same vaccine delivered IM using the Medical International Technologies Inc. (MIT) compressed air vaccine delivery system (Med-Jet H4).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Observer-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jet injector (Active Comparator): 40 participants will receive Fluviral influenza vaccine using the Med-Jet H4
  Interventions: Biological: Fluviral influenza vaccine
- IM injection (pre-filled syringe) (Active Comparator): 20 participants will receive Fluviral influenza vaccine using pre-filled syringes for time-motion comparison to Med-Jet H4
  Interventions: Biological: Fluviral influenza vaccine
- IM injection (multi-dose vial) (Active Comparator): 20 participants will receive Fluviral influenza vaccine using a multi-dose vial for time-motion comparison to Med-Jet H4
  Interventions: Biological: Fluviral influenza vaccine

INTERVENTIONS:
Biological: Fluviral influenza vaccine — Influenza vaccine (Fluviral) given via Med-Jet H4 or IM injection

SUMMARY:
80 subjects (healthy adults) will be randomized to receive the seasonal flu vaccine either by needle & syringe or by the MIT needle-free injector (Med-Jet MIT H4™ & Disposable Cartridge). The study will be conducted after the normal flu season has passed (ie: March-April). Half of those randomized to standard vaccination (n=20) will receive vaccine drawn from a multi-dose vial while the other half (n=20) will receive vaccine drawn from a single use vial. The same vaccine as the multi-dose vial will be delivered to the other half of the subjects (n=40) using the MIT injector. How long it takes to prepare and deliver the vaccines will be assessed (a time-motion study). Subject acceptance before and after injection will be assessed as well as local and systemic side effects. Standard serologic measures of immune response to flu vaccination (ie: antibodies) will determine whether the Med-Jet H4 injector induces the same kind of immune response as needle & syringe delivery.

DETAILED DESCRIPTION:
Eighty healthy adults (18-49 years of age) will be randomized 1:1 to receive:

* A single dose of trivalent inactivated influenza vaccine (TIV: Fluviral™: 0.5mL IM)

  * Half will receive the vaccine using a pre-filled syringe
  * Half will receive the vaccine using a multi-dose vial
* Or,the same vaccine delivered IM using the Medical International Technologies Inc. (MIT) compressed air vaccine delivery system (Med-Jet MIT H4 & Disposable Cartridge).

Primary study outcomes will be i) safety (local and systemic reactions) followed for 21 days and ii) immunogenicity at 21 days using the standard serologic assays (eg: hemaggultination inhibition (HI) and microneutralization (MN)).

Secondary outcomes will be time-motion analyses of vaccine preparation and administration to assess possible time-saving associated with Med-Jet H4 delivery.

Although full blinding of the study is not possible give the very different vaccine delivery methods, all safety assessments and immunological parameters will be collected by nurses/technicians blinded to group assignment (ie: observer blind).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults
* 18 to 49 years of age
* body mass index (BMI) of ≥ 18 kg/m2 and ≤ 32 kg/m2
* Must be accessible by phone on a consistent basis and be available for the D21 blood draw

Exclusion Criteria:

* Any influenza vaccine during the 2016-2017 season
* significant acute or chronic, uncontrolled medical or neuropsychiatric illness
* confirmed or suspected immunosuppressive condition or immunodeficiency
* history of autoimmune disease, cancer, or treatment for cancer within 3 years of study vaccine administration
* Receipt of any investigational or non-registered product within 30 days prior to study enrolment
* receipt of systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent, for more than 7 consecutive days or for 10 or more days in total within 1 month of vaccine administration
* any other cytotoxic or immunosuppressant drug or any globulin preparation within 3 months of vaccination
* blood transfusion within 90 days of study vaccination
* Although there is no known danger from influenza vaccination during pregnancy, pregnant women will be excluded since the efficacy of the Med-Jet delivery system is not yet known
* known drug or alcohol abuse will also be excluded.

Temporary Contraindications Following the resolution, in the opinion of the Investigator, of the following temporary conditions that constitute contraindications to administration of study vaccine, subjects may be enrolled in the study:

* Temperature ≥ 38.0 ºC within 24 hours prior to randomization.
* Acute cold symptoms such as upper respiratory tract infection symptoms, with or without fever, which typically resolve in 48 to 72 hours prior to randomization.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Local and systemic effects will be measured after vaccination | 0 - 21 days
  Solicited and unsolicited local and systemic adverse events will be collected between day 0-3 by phone and day 4-21 by diary after influenza vaccine (TIV) delivered by jet-injector or by standard needle.

SECONDARY OUTCOMES:
Time to administer vaccine by jet-injector or standard needle will be measured | Day 0 (day of immunization)
  Each component of the vaccination process using either the jet-injector or a standard needle will be measured (time-motion study) to determine which method is faster
Immunogenicity of influenza vaccine given by needle or jet injector | Day 0 (day of immunization) and day 21
  Standard serologic assays will be performed on serum obtained on day 0 (day of injection) and day 21 to measure hemagglutination inhibition and microneutralization titres in subjects who received the vaccine by either standard needle or jet injector.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Ward, MD, Principal Investigator — Research Institute of the McGill University Helath Centre
Locations (1):
- McGill University Health Centre Vaccine Study Centre, Pierrefonds, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shapiro JR, Hodgins B, Hendin HE, Patel A, Menassa K, Menassa C, Menassa M, Pereira JA, Ward BJ. Needle-free delivery of influenza vaccine using the Med-Jet(R) H4 is efficient and elicits the same humoral and cellular responses as standard IM injection: A randomized trial. Vaccine. 2019 Feb 28;37(10):1332-1339. doi: 10.1016/j.vaccine.2019.01.039. Epub 2019 Jan 29. PMID 30709725